CLINICAL TRIAL: NCT06982066
Title: Improving Health-Related Quality of Life Communication Between AYA Oncology Patients and Clinicians: A Patient-Centered Intervention
Brief Title: Improving Communication Between AYA Oncology Patients and Clinicians: A Patient-Centered Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-081; K08CA286736 (NIH)
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Pediatric Cancer; Adolescent and Young Adult Cancer
Keywords: adolescent young adult; sexual health communication; cancer; patient provider communication; sexual and reproductive health
MeSH Terms: conditions — Neoplasms; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ReSPECT (Experimental): Aims 2 and 3 involve a single-arm cohort study of the ReSPECT intervention using a pre-post design. Enrolled participants will complete a survey at baseline, immediately after intervention use, and at 2 months from study enrollment. All participants will also be invited to participate in a brief interview immediately after intervention use.
  Interventions: Behavioral: ReSPECT

INTERVENTIONS:
Behavioral: ReSPECT — ReSPECT is an interactive, web-based digital platform that integrates (1) an AYA-centered pre-visit questionnaire (PVQ) that will discretely alert clinicians to relevant SRH questions/concerns, (2) targeted patient education on PVQ selections, and (3) clinician-centered guidance for addressing SRH issues. At enrollment, all participants will complete a baseline survey (T1). AYAs will have access to the ReSPECT digital platform and will receive the first prompt to complete the PVQ 3-5 days before their next clinic appointment. Once completed, AYAs will receive an email/text with a link to tailored information based on their PVQ selections for review. Clinicians will receive an email with a link to the patient's PVQ results on the ReSPECT platform along with clinical management recommendations. All participants will complete a brief virtual survey (T2) and interview within 48 hours of the first postintervention clinic visit and a follow-up survey 2 months after study enrollment (T3).

SUMMARY:
The overarching goal is to develop and demonstrate proof-of-concept of ReSPECT (Reproductive and Sexual Health Patient Education and Communication Tool), a multi-modal communication intervention to improve adolescent and young adult (AYA)- clinician sexual and reproductive health (SRH) communication in the outpatient oncology clinic setting.

DETAILED DESCRIPTION:
To improve sexual and reproductive health communication between adolescent and young adult oncology patients and their clinicians, the Investigator will be developing and testing proof-of-concept of a novel web-based intervention called ReSPECT (Reproductive and Sexual health Patient Education and Communication Tool). The overarching goal of this proposal is to develop and pilot test a patient-centered approach to improve sexual and reproductive health communication during cancer care.

Prior to the clinical trial, Aim 1 of this study will develop and refine ReSPECT by integrating feedback from AYAs and pediatric oncology clinicians on individual intervention components followed by additional feedback collected through cognitive debriefing. Once Aim 1 is completed, the intervention will be ready for proof-of-concept testing.

Aims 2 and 3 involve a single-arm cohort study of the ReSPECT intervention using a pre-post design. Enrolled participants will complete a survey at baseline, immediately after intervention use, and at 2 months from study enrollment. All participants will also be invited to participate in a brief interview immediately after intervention use.

ELIGIBILITY:
Inclusion Criteria

Adolescent and Young Adult Oncology Patients

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Be aged 15-25 years old at time of enrollment.
2. Have a cancer diagnosis and currently be on cancer-directed therapy with at least one of the following:

   1. Chemotherapy: any anticancer drug to treat the cancer diagnosis, including immunotherapy.
   2. Radiotherapy: any radiotherapy to treat the cancer diagnosis.
   3. Surgery: any surgery to remove cancer including partial of total resections. Biopsies are not considered surgery.
3. Be greater than or equal to 2 months from diagnosis/initiation of therapy, whichever occurred later.
4. Be able to speak and read English
5. Have permission to participate from a member of the patient's primary oncology team.
6. Provision to sign and date the consent/assent form.
7. Active study participation of primary oncology clinician
8. Patient must have primary oncology care at Connecticut Children's Center for Cancer & Blood Disorders of Children's Hospital Los Angeles Cancer & Blood Disease Institute

Exclusion Criteria

An individual who meets and of the following criteria will be excluded from participation in this study:

1. Not currently on cancer-directed therapy.
2. Unable to speak and read English.
3. Insufficient cognitive functioning to complete study measures (as determined by a member of the patient's primary oncology team)

Pediatric Oncology Clinicians

1. Be a pediatric oncology physician, clinical fellow, or advanced practice provider (including nurse practitioners and physician assistants) that provides clinical care for AYA patients with cancer

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2029-03-15 (Estimated); Study Completion 2029-06-29 (Estimated)

PRIMARY OUTCOMES:
Feasibility of implementing the ReSPECT intervention. | 2 months
  Feasibility will be based on patient recruitment and completion of the intervention. The intervention will be considered feasible if AYA recruitment is greater than or equal to 60% and if greater than or equal to 80% of consented AYAs complete the intervention (retention). Intervention completion will be defined as AYA completion of the pre-visit questionnaire and post-intervention survey.
Acceptability of the ReSPECT intervention. | 2 months
  The intervention will be considered acceptable if greater than or equal to 70% of AYA and clinician participants rate ReSPECT as acceptable (average score of 4 or higher) on the Lyon Satisfaction Questionnaire, adapted for this study, which includes a 10-item satisfaction questionnaire where 1 is strongly disagree and 5 is strongly agree. Subjects will report via survey after the healthcare visit.
Usability of the ReSPECT intervention. | 2 months
  The intervention will be considered usable/sustainable if greater than or equal to 70% of AYA and clinician participants rate ReSPECT as usable (average score of 4 or higher) on the Usability/Sustainability of Intervention Scale, adapted for this study, on a 4-item usability questionnaire where 1 is strongly disagree and 5 is completely agree. Subjects will report via survey after the healthcare visit.
Perceived utility of the ReSPECT intervention. | 2 months
  Through qualitative interviews, participants will be asked for their perceptions on the impact of ReSPECT in promoting SRH communication in the outpatient clinic setting.

SECONDARY OUTCOMES:
Comparison of patient reported SRH communication before and after intervention implementation. | 2 months
  Comparison of pre- and post- intervention percentage of patients reporting that their clinician talked to them about a SRH topic during the most recent clinic visit. Subjects will report via survey (yes/no) at baseline and after their healthcare visit.
Comparison of clinician reported SRH communication before and after intervention implementation. | 2 months
  Comparison of pre- and post- intervention percentage of clinicians reporting that they talked to their AYA patient about a SRH topic during the most recent clinic visit. Subjects will report (yes/no) via survey at baseline and after the healthcare visit.
Comparison of patient self-efficacy in discussing SRH topics with their oncology clinician before and after intervention implementation. | 2 months
  Comparison of pre- and post- intervention patient report of confidence in talking to their oncology clinician about SRH. Patients will complete a multi-item questionnaire adapted for this study on confidence where 0 is "not at all confident" and 10 is "extremely confident." Subjects will report via survey at baseline and after the healthcare visit.
Comparison of clinician of self-efficacy in discussing SRH topics with their AYA patient before and after intervention implementation. | 2 months
  Comparison of pre- and post- intervention clinician report of confidence in talking to their AYA clinician about SRH. Patients will complete a multi-item questionnaire adapted for this study on confidence where 0 is "not at all confident" and 10 is "extremely confident." Subjects will report via survey at baseline and after the healthcare visit.
Comparison of patient- reported outcome expectancies related to discussing SRH topics with their oncology clinician before and after intervention implementation. | 2 months
  Comparison of pre- and post- intervention patient report of perceived benefit of discussing SRH with their clinician. Patients will complete a 6-item questionnaire adapted for this study on perceived benefit where 0 is "not at all" and 10 is "very much." Subjects will report via survey at baseline and after the healthcare visit.
Intervention impact on decision-making. | 2 months
  The proportion of patients that report the intervention helped them get the information that they needed to make informed decisions about SRH. Subjects will report (yes/no) via survey after their healthcare visit.
Comparison of patient-reported distress/bother by SRH-related questions or concerns before and after the intervention. | 2 months
  Comparison of pre- and post- intervention rating of distress/bother by SRH-related questions or concerns. Patients will complete a single item scale on the degree of bother on the Distress/Bother Scale where 1 is "Not at all bothersome" and 4 is "Bothers me a lot". Subjects will report via survey at baseline and after the healthcare visit.
Comparison of patient-reported engagement in sexual health risk behaviors before and after the intervention. | 2 months
  Comparison of patient-reported engagement in sexual health risk behaviors pre- and post- intervention implementation. Patients will complete a study-specific survey consisting of several questions about engagement in sexual health risk behaviors (yes/no and nominal). Subjects will report via survey at baseline and after the healthcare visit.
Comparison of patient-reported therapeutic alliance before and after the intervention. | 2 months
  Comparison of patient-reported therapeutic alliance with primary oncology clinician pre- and post- intervention implementation. Patients will complete 16 items on The Human Connection Scale (4-point scale). Subjects will report via survey at baseline and after the healthcare visit.

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Frederick, MD, MPH, Principal Investigator — nfrederick@connecticutchildrens.org
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States